CLINICAL TRIAL: NCT07222735
Title: Hypofractionated Radiation in Combination With B7-H3-CAR T Cells for Pediatric Patients With Relapsed/Refractory Sarcomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD3CAR; NCI-2025-07135 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Sarcoma; Childhood Osteosarcoma; Childhood Rhabdomyosarcoma; Childhood Soft Tissue Sarcoma; Ewing Sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Ewing | interventions — fludarabine; Cyclophosphamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RAD3CAR Treatment (Experimental): Peripheral blood mononuclear cells (PBMC) will be collected by autologous apheresis.
  Treatment will include HFRT to at least one site of disease, administered in parallel with a single course of lymphodepleting chemotherapy (fludarabine/cyclophosphamide) and followed by CAR T cell infusion.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: B7-H3-CAR T Cells; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Fludarabine — Intravenously on day -5, -4, -3 and -2
Drug: Cyclophosphamide — Intravenously on day -3, -2
Drug: B7-H3-CAR T Cells — Intravenously on day 0
Radiation: Radiation Therapy — 5 or 8 treatment sessions (fractions), scheduled to complete on Day -2

SUMMARY:
RAD3CAR is a phase I study designed to evaluatethe safety of B7-H3-CAR T cells and lymphodepletion in combination with hypofractionated radiation therapy.

Primary objective:

- To evaluate the safety of B7-H3-CAR T cell therapy after priming with hypofractionated radiation therapy (HFRT) and lymphodepleting chemotherapy in patients ≤ 21 years of age with relapsed/refractory B7-H3+ sarcomas.

Secondary objectives:

* To describe the antitumor activity of B7-H3-CAR T cells in combination with HFRT
* To determine if B7-H3-CAR T cells traffic to tumor sites after combination treatment with HFRT

DETAILED DESCRIPTION:
This study is a phase I study designed to describe the safety of B7-H3-CAR T cells and lymphodepletion in combination with hypofractionated radiation therapy for the treatment of pediatric patients with B7-H3+ sarcoma.

The study will contain two-part eligibility criterion: one to proceed with autologous apheresis and manufacturing of CAR T cells, and a second to proceed with CAR T cell treatment.

The primary intervention is the administration of autologous B7-H3-CAR T cells, after priming with HFRT and administration of lymphodepleting chemotherapy. Peripheral blood mononuclear cells (PBMC) will be collected by autologous apheresis. Treatment will include HFRT to at least one site of disease, administered in parallel with a single course of lymphodepleting chemotherapy (fludarabine/cyclophosphamide) and followed by CAR T cell infusion. Participants are evaluated for a post-treatment tumor biopsy and may choose to be evaluated for a pre-treatment tumor biopsy. Participants who meet specified criteria will be eligible for optional additional treatment courses.

ELIGIBILITY:
INCLUSION CRITERIA

*a previously collected, autologous leukapheresis product can be used for T cell production

Collection and manufacturing eligibility

* Age ≤ 21 years old
* B7-H3+ sarcoma; B7-H3 expression will be evaluated by standard immunohistochemistry (IHC) using any previously obtained biopsy; a tumor is considered B7-H3 positive with a H score greater than or equal to 100

  * Osteosarcoma
  * Ewing Sarcoma
  * Rhabdomyosarcoma Non-rhabdomyosarcoma soft tissue sarcomas
* Evidence of relapsed (cancer that has completely responded [i.e., no evidence of disease using standard imaging modalities] to first-line therapy but has recurred for the first or subsequent time); or refractory (cancer that does not respond completely to treatment; cancer may be resistant at the beginning or may become resistant during treatment) disease after standard first-line therapy
* Evaluable disease with presence of at least one lesion amenable to hypofractionated radiation therapy

  * For dose expansion cohort: participants must also have additional evaluable disease beyond planned radiation field
* Estimated life expectancy of > 12 weeks
* Karnofsky or Lansky (age-dependent) performance score ≥ 60

  * Participants with mobility limitations due to prior surgical intervention (i.e., amputation) but who are up in wheelchair or with other assistive devices will be considered ambulatory for the purpose of performance score determination
* For females of child-bearing age:

  * Not pregnant with negative serum pregnancy test within 7 days prior to enrollment
  * Not lactating with intent to breastfeed
* Participants must be eligible to undergo autologous apheresis or have an available previously collected autologous apheresis product

Treatment eligibility

* Age ≤ 21 years old at the time of manufacturing
* B7-H3+ sarcoma
* Evidence of relapsed or refractory disease after standard first-line therapy
* Evaluable disease with the presence of at least one lesion amenable to hypofractionated radiation therapy

  • For dose expansion cohort: participants must also have additional evaluable disease beyond the planned radiation field
* Estimated life expectancy of > 8 weeks
* Karnofsky or Lansky (age-dependent) performance score ≥ 60

  • Participants with mobility limitations due to prior surgical intervention (i.e., amputation) but who are up in wheelchair or with other assistive device will be considered ambulatory for purpose of performance score determination.
* Adequate cardiac function defined by echocardiogram with left ventricular ejection fraction ≥ 50%
* Adequate renal function as defined by not exceeding the maximum serum creatinine listed below by age:

  * 1 to <2 years: 0.6
  * 2 to <6 years: 0.8
  * 6 to <10 years: 1
  * 10 to <13 years: 1.2
  * 13 to <16 years: male 1.5, female 1.4
  * ≥ 16 years: male 1.7, female 1.4
* Adequate pulmonary function defined as pulse oximetry ≥ 92% on room air
* Total Bilirubin ≤3 times the upper limit of normal for age, except in subjects with Gilbert's syndrome
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤5 times the upper limit of normal for age
* Hemoglobin ≥ 7g/dL (can be transfused)
* Platelet count ≥ 50,000/μL (can be transfused)
* Absolute neutrophil count (ANC) ≥ 1000/μL
* Has recovered from all NCI CTAE grade III-IV, non-hematologic acute toxicities from prior therapy
* For females of child-bearing age:

  * Not pregnant with negative serum pregnancy test within 7 days prior to enrollment
  * Not lactating with intent to breastfeed
* If sexually active, agreement to use contraception until 3 months after T cell infusion

EXCLUSION CRITERIA

Collection and manufacturing eligibility

* Known primary immunodeficiency
* Known HIV positivity
* Severe, uncontrolled intercurrent bacterial, viral, or fungal infection
* Known active malignancy other than the B7-H3+ sarcoma being treated on study
* Rapidly progressive disease (as assessed by the study PIs, with consideration for proximity to critical structures)
* Presence of intracranial or spinal cord disease
* Known underlying medical condition(s) for which, in the investigator's opinion, participation in this trial would not be in the best interest of the participant (e.g., compromises the health of the subject) or that could prevent, limit, or confound protocol assessments
* Known severe hypersensitivity to corn starch or hydroxyethyl starch

Treatment eligibility

* Known primary immunodeficiency
* Known HIV positivity
* Severe, uncontrolled intercurrent bacterial, viral, or fungal infection
* Known active malignancy other than the B7-H3+ sarcoma being treated on study
* Receiving systemic steroid therapy exceeding the equivalent of 0.5 mg/kg/day of methylprednisolone, < 7 days prior to CAR T cell infusion
* Receiving systemic therapy < 14 days prior to start of protocol therapy, which will interfere with the activity of the CAR product (in the opinion of the study PIs)
* Received radiation therapy within the 4 weeks prior to start of protocol therapy
* Rapidly progressive disease (as assessed by the study PIs, with consideration for proximity to critical structures)
* Presence of intracranial or spinal cord disease
* Known underlying medical condition(s) for which, in the investigator's opinion, participation in this trial would not be in the best interest of the participant (e.g., compromises the health of the subject) or that could prevent, limit, or confound protocol assessments
* Known severe hypersensitivity to corn starch or hydroxyethyl starch

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2030-11-05 (Estimated); Study Completion 2031-11-05 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) rate | up to 4 weeks after CAR T cell infusion
  Proportion of evaluable participants experiencing DLTs
Incidence of adverse events (AEs) | up to 4 weeks after CAR T cell infusion
  AEs will be assessed and graded using CTCAE v5.0, except for cytokine release syndrome (CRS) and immune effector cell associated neurotoxicity syndrome (ICANS), which will be graded according to ASTCT consensus guidelines. AEs will be summarized and reported descriptively

SECONDARY OUTCOMES:
Clinical antitumor activity | 4-12 weeks after CAR T cell infusion
  Best overall response after treatment as determined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, and if applicable bone marrow evaluation
B7-H3-CAR T cell trafficking to tumor sites | 2 weeks after CAR T cell infusion
  Evaluate for the presence of B7-H3-CAR T cells in post-treatment tumor biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Epperly, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org